CLINICAL TRIAL: NCT03890614
Title: Novel 3D Hematological Malignancy Organoid Platform to Study Disease Biology and Perform Chemosensitivity Assays for Patient-Specific Care
Brief Title: Novel 3D Hematological Malignancy Organoid to Study Disease Biology and Chemosensitivity
Acronym: Organoid
Status: Recruiting | Type: Observational
Sponsor: Wake Forest University Health Sciences (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Other Study IDs: IRB00057612; Crowdcare Foundation (Other Grant/Funding Number: GTS 47809); Pilot Fund (Other: CTSI); P30CA012197 (NIH); WFBCCC26A19 (Other: WFCCC)
Record Dates: First submitted 2019-03-18; First posted 2019-03-26 (Actual); Last update posted 2025-03-04 (Actual); Status verified 2025-03

CONDITIONS: Hematologic Malignancy
Keywords: 3D organoid technique
MeSH Terms: conditions — Hematologic Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Bone marrow
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Ancillary-Correlative - Creation of three-dimensional myeloma organoids using marrow aspirates — Bone marrow aspirates will be collected from participants with hematologic malignancy being evaluated for relapsed disease to create three-dimensional constructs using a three-dimensional bioprinting methodology for automated organoid biofabrication.

SUMMARY:
The objective of this project is to compare chemosensitivity between chemotherapy combinations in bone marrow aspirates using 3D organoid models. The investigators overarching hypothesis is that 3D organoids are ideal to test chemosensitivity in real time, to provide personalized medicine and guidance in the setting of relapsed hematologic malignancy and potentially other cancers.

DETAILED DESCRIPTION:
Optimize the novel 3D organoid technique already used to recreate myeloma tumors in the Regenerative Medicine laboratory.

Optimize cell viability of myeloma organoids to extend available time in culture by screening cell culture media cytokines and 3D extracellular matrix composition (current environment is able to maintain cells alive for up to 5-7 days to allow testing).

Evaluate myeloma tumor markers at different time points of organoid life to confirm accurate tumor representation, identify genetic expression characteristics, unique mutations, and tumor-stroma interaction. This will give information of the tumor characteristics to learn about tumor biology and correlate with responses.

Evaluate chemosensitivity on patient derived 3D organoids. Using myeloma patients marrow aspirate, evaluate live/kill rates of myeloma cells after being exposed to established regimen combinations after 24 and 36 hours of exposure at pre-determined concentrations.

Using patient samples, evaluate differences in gene expression and cell markers of the myeloma cells that remained alive after chemotherapy exposure to better understand mechanisms of resistance.

Validate the predictive value of the 3D organoid chemobiogram results compared with retrospective data of the donor s responses to the treatment used at that time point. This will compare in vivo/ex vivo responses and facilitate future personalized medicine. Chemobiogram is the report on chemosensitivity from the combinations tested much like an antibiogram.

ELIGIBILITY:
Inclusion Criteria:

* Patients with suspected or confirmed hematologic malignancy undergoing a bone marrow biopsy as part of their care.
* The ability to understand and willingness to sign an IRB approved informed consent document.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Hematologic malignancy patients undergoing transplant.
Sampling Method: Probability Sample
Enrollment: 70 (Estimated)
Dates: Start 2019-05-16 (Actual); Primary Completion 2026-02 (Estimated); Study Completion 2026-02 (Estimated)

PRIMARY OUTCOMES:
Proportion of Live/Dead Myeloma Cells Using Bioprinting Technology | Up to 5 days
  Bone marrow aspirates (around 3-7 ml) will be collected from patients with hematologic malignancy being evaluated for relapsed disease. The samples will be used to create 3D organoid constructs using a 3D bioprinting technology for automated organoid biofabrication using hyaluronic acid and gelatin-based hydrogel. The 3D organoid constructs allow extended time to simulate the protective environment cancer cells use to survive in bone marrow. Organoids will be assessed at 1, 3, and 5 days for viability of myeloma cells. Based on live/dead cells using fluorescent imaging, the hydrogel composition will be modified to allow the optimal media for cell survival ex vivo.
Tumor-Stroma Interactions | Up to 5 days
  To assess the interaction of myeloma cells with stromal cells in a 3D organoid model, plasma and myeloma cells will be labeled using differing colors of Vybrant Multicolor Cell Labeling Kit to allow visualization of the cells' nuceli. By confocal microscope, slides will be evaluated for Vybrant-labeled hematologic malignant cells or healthy plasma cells (different colors) to identify preferential cell interactions. These aspects of tumor interaction with its stromal microenvironment will provide critical knowledge to better understand its biology.

SECONDARY OUTCOMES:
Number of Reduced Hematologic Malignant Myeloma Cells | Up to 3 days
  After 24 hours of incubation, chemotherapy agents will be added at prepared concentrations that fall within the prescribed therapeutic ranges. A maximum of 15 combinations for each donor will be allowed for testing after which the efficacy of the treatments will be assessed qualitatively (live/dead straining) and quantitatively and quantitatively (automated segmentation and quantification of live/dead staining, mitochondrial metabolism/ATP activity, and ratio of Annexin V staining versus Ki67 staining [apoptosis versus proliferation]). These metrics will capture the reduction in hematologic malignant cell population.
Comparison of Cell Viability | 24 and 36 hours
  Using myeloma patients' marrow aspirate, evaluate live/kill rates of myeloma cells after being exposed to established regimen combinations after 24 and 36 hours of exposure at pre-determined concentrations.
Organoid Responses Compared to Clinical Response | Up to 3 months
  The response to each chemotherapy agent from obtained three-dimensional organoids will be compared to actual clinical responses of each participant through retrospective chart review to obtain regimen used to treat disease and the level of measurable disease in serum at different time points of treatment. The time points would include time of marrow biopsy, after 2 cycles of treatment and after 4 cycles of treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Timothy Pardee, MD, PhD, Principal Investigator — Wake Forest University Health Sciences
Locations (1):
- Wake Forest Baptist Comprehensive Cancer Center, Winston-Salem, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No